CLINICAL TRIAL: NCT05633069
Title: Interest of Instantaneous Fluctuations of Pupillary Diameter for Pain Evaluation in Intensive Care Sedated Patients.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN412014/CHUSTE
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Intubation Complication
Keywords: Fluctuation of pupillary diameter; Variation coefficient of pupillary diameter; Pain monitoring; Behavioral Pain Scale; Videopupillometer; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring orotracheal intubation or tracheostomy: Patients hospitalized in the surgical Intensive Care Unit (ICU) of the University Hospital of Saint-Etienne between September 2015 and August 2016 for medical-surgical pathologies, requiring orotracheal intubation or tracheostomy, and presenting on the day of recording a Riker sedation score of 3 or 4 will be included.
  Datas analysed by medical records.
  Interventions: Other: Datas analysed by medical records

INTERVENTIONS:
Other: Datas analysed by medical records — Datas analysed by medical records : pupillary parameters: pupillary diameter and pupillary diameter variation. heart rate, the blood pressure, the Behavioral Pain Scale (BPS) pain score before and during painful procedures.
  The pupillary parameters were recorded with the AlgiScan® pupillometer (iDMed, Marseille, France), which allows the recording of Pupillary Diameter (PD) variations at the patient's bed at a sampling frequency of 67 hertz.

SUMMARY:
New pain assessment parameter, called the Variation Coefficient of Pupillary Diameter (VCPD) described. This parameter allows evaluating the pain of patients during uterine contractions in obstetrical labor, and postoperatively in recovery room.

This parameter also allows evaluating the level of pain in Intensive Care Unit (ICU), in intubated or tracheotomized patients moderately sedated (Riker score 3 or 4).

DETAILED DESCRIPTION:
This study propose to recalculate the Variation Coefficient of Pupillary Diameter (VCPD) from pupil recordings performed in the Intensive Care Unit (ICU) in 2015-2016 and kept in the patients' records. From there, the Variation Coefficient of Pupillary Diameter (VCPD) will compare to the Behavioral Pain Scale (BPS), considered the gold standard pain assessment

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in the surgical Intensive Care Unit (ICU) of the University Hospital of Saint-Etienne between September 2015 and August 2016 for medical-surgical pathologies
* requiring orotracheal intubation or tracheostomy
* and presenting a Riker sedation score of 3 or 4.

Exclusion Criteria:

* cerebral palsy
* curarization
* paraplegia or tetraplegia
* intensive care neuromyopathy
* ocular pathology
* history of severe dysautonomic disease that could influence the evaluation of the Behavioral Pain Scale (BPS) or Variation Coefficient of Pupillary Diameter (VCPD) score
* receiving antiarrhythmic treatment that could make the interpretation of the results difficult
* on metoclopramide, droperidol, clonidine, or dexmedetomidine, which are known to alter the pupil dilation reflex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the surgical Intensive Care Unit (ICU) of the University Hospital of Saint-Etienne between September 2015 and August 2016 for medical-surgical pathologies, requiring orotracheal intubation or tracheostomy, and presenting on the day of recording a Riker sedation score of 3 or 4 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Correlation between fluctuations in Pupillary Diameter (PD), as assessed by the Variation Coefficient of Pupillary Diameter (VCPD) and the level of pain. | Months: 1
  Variation Coefficient of Pupillary Diameter (VCPD) calculate from continuous pupil recordings during tracheal aspirations, considered as a painful procedure.
  The nurse in charge of the patient scored the Riker sedation score before endotracheal suctioning and the pain level estimated by the Behavioral Pain Scale (BPS) scale before and during endotracheal suctioning.

CONTACTS AND LOCATIONS:
Overall Officials: David CHARIER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No